CLINICAL TRIAL: NCT00212212
Title: Human Selenium Nutritional Requirement and Biomarkers in Health and Disease
Brief Title: Selenium Supplementation of Patients With Cirrhosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funds to complete study.
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, RBurk, M.D., Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: DK58763; R01DK058763 (NIH); R01DK058763-06 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-21 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Cirrhosis
Keywords: selenium supplements; selenate; selenomethionine; biomarkers; plasma selenium concentration; plasma glutathione peroxidase; selenoprotein P
MeSH Terms: conditions — Fibrosis | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 200 µg selenium as selenate
  Interventions: Dietary Supplement: selenium
- 2 (Experimental): 400 µg selenium as selenate
  Interventions: Dietary Supplement: selenium
- 3 (Experimental): 200 µg selenium as selenomethionine
  Interventions: Dietary Supplement: selenium
- 4 (Placebo Comparator): placebo tablet
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: selenium — 200 µg selenium as selenate
  Arms: 1
Dietary Supplement: selenium — 400 µg selenium as selenate
  Arms: 2
Dietary Supplement: selenium — 200 µg selenium as selenomethionine
  Arms: 3
Dietary Supplement: placebo — placebo tablet
  Arms: 4

SUMMARY:
This study is being conducted to determine if patients with cirrhosis (liver disease) are selenium deficient. The effect of supplementation with two chemical forms of selenium on plasma selenium biomarkers will be determined and correlated with the severity of the liver disease.

DETAILED DESCRIPTION:
Selenium is an essential nutrient that plays a role in oxidant defense, among other functions. There is much interest in the role selenium may play in several disease processes. It is possible that certain diseases result in selenium deficiency because of the form of selenium taken in the normal diet.

We propose to measure the selenium biomarkers associated with supplemental intakes of 200 or 400 µg of selenium per day in the chemical form selenate, or with supplemental intake of 200 µg selenium as selenomethionine. 144 patients with cirrhosis will be randomized to one of 4 treatment groups, including a placebo. After treatement for 4 weeks, all participants will receive 400 µg of selenium per day as selenate for 4 weeks. Blood will be measured initially and at 4 and 8 weeks. Selenium, selenoprotein P and glutathione peroxidase will be measured in the plasma.

ELIGIBILITY:
Inclusion Criteria:

* adults with cirrhosis

Exclusion Criteria:

* Pregnancy or planning a pregnancy
* Selenium supplements of 25 µg or more within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Plasma selenium biomarkers | 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F Burk, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States